CLINICAL TRIAL: NCT07143591
Title: Outcome of Supraventricular Tachycardia in Children Admitted to Assuit University Children Hospital
Brief Title: Outcome of SVT in Children Admitted to AUCH
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sameh Mounir Moussa Soliman, Pediatric resident, Assiut University
Other Study IDs: Outcome of SVT in children
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Supraventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Supraventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Not found — No intervention

SUMMARY:
The aim of the study is to:

. Assess the outcome of Supraventricular tachycardia , the most effective acute and long-term management strategies and recurrence rates of SVT .

DETAILED DESCRIPTION:
Supraventricular tachycardia (SVT) is the most common symptomatic arrhythmia in the pediatric population, characterized by an abnormally rapid heart rate that originates above the ventricles-typically involving the atrial tissue or the atrioventricular (AV) node. It affects approximately

1 in 500 children. Clinical presentation varies by age. Infants may present with poor feeding, vomiting, irritability, lethargy, diaphoresis, or syncope, and may show signs of congestive heart failure if undiagnosed. Older children may report palpitations, chest discomfort, dizziness, shortness of breath, or syncope . Initial management of pediatric SVT follows the ABCDE approach (Airway, Breathing, Circulation, Disability, Exposure) to assess stability. In stable patients, treatment begins with VAGAL maneuvers, followed by ADENOSINE (0.1 mg/kg IV bolus), if needed. If adenosine fails, antiarrhythmic drugs such as β-blockers, flecainide, or amiodarone may be used. In unstable SVT, immediate synchronized cardioversion (0.5-2 J/kg) is indicated. For recurrent SVT, long-term management may include the FLEA approach: Flecainide, Lifestyle modification, Electrophysiologic study, and Ablation. Paroxysmal supraventricular tachycardias (SVTs) are considered benign if the electrocardiogram in sinus rhythm is normal, but their occurrence in children/teenagers is often associated with anxiety in parents, children and their doctors, and sometimes with embarrassing and invalidating symptoms.Invasive evaluation of tachycardia is rarely indicated for several reasons, including misdiagnosis or fear of hospitalization. Frequently, children/teenagers who complain of palpitations or tachycardia are only considered to be anxious, and for several months or years a false diagnosis of sinus tachycardia is given. It is important to provide education and counseling to patients and their families, including information about the condition, treatment options, potential complications, and psychological support. Outcomes of Supraventricular Tachycardia (SVT) in Children, Most children recover fully, either by outgrowing SVT or with curative ablation. Long-term survival is excellent, with no reduction in life expectancy in isolated SVT.. About 30-50% of infants outgrow SVT by age 1-2 . 70-85% of children do well with medications . <5% of infants with untreated SVT may develop heart failure . <1% are at risk of serious events like sudden death . Over 95% grow and develop normally. In this study, the outcome of SVT in pediatrics is assessed including the clinical and electrophysiological data , the most effective acute and long-term management and recurrence rates.

ELIGIBILITY:
Inclusion Criteria:

* Children aged greater than 1 month and up to 18 years
* Diagnosis of supraventricular tachycardia (SVT) based on:
* Clinical presentation
* Electrocardiogram (ECG) findings

Exclusion Criteria:

* Presence of structural heart disease
* Incomplete clinical data
* Lost to follow-up during the study period

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All with the required criteria
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Outcome of Supraventricular tachycardia in children and recurrence rates | Baseline
  Assess the outcome of Supraventricular tachycardia , the most effective acute and long-term management strategies and recurrence rates of SVT .

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hafeez Y, Quintanilla Rodriguez BS, Ahmed I, Grossman SA. Paroxysmal Supraventricular Tachycardia. 2024 Feb 28. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK507699/ PMID 29939521
- [Background] Nasir M, Sturts A, Sturts A. Common Types of Supraventricular Tachycardia: Diagnosis and Management. Am Fam Physician. 2023 Jun;107(6):631-641. PMID 37327167